CLINICAL TRIAL: NCT03661216
Title: A Prospective, Double-Blind, Randomized, Placebo-Controlled, Cross-Over Study With Nephure™, an Orally Administered Oxalate Reducing Enzyme
Brief Title: Evaluation of Nephure™, and the Reduction of Dietary Oxalate, in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Captozyme, Inc. (Industry)
Responsible Party: Principal Investigator, Donald Burkindine, D.O., Principal Investigator, QPS-Qualitix
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 95318
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, cross-over study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double (participant and investigator) and outcomes assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 3g of non-GMO maltodextrin
  Interventions: Other: Placebo
- Nephure (Active Comparator): 3g of Nephure
  Interventions: Dietary Supplement: Nephure Oxalate-reducing Enzyme

INTERVENTIONS:
Dietary Supplement: Nephure Oxalate-reducing Enzyme — 3g of Nephure is mixed with 8oz of water and ingested with breakfast, lunch and dinner.
  Arms: Nephure
Other: Placebo — 3g of non-GMO maltodextrin is mixed with 8oz of water and ingested with breakfast, lunch and dinner.
  Arms: Placebo

SUMMARY:
The purpose of this double-blind study is to determine the effect of reducing oxalates in the diet of healthy volunteers by using Nephure, an oxalate-reducing enzyme, as compared to placebo.

DETAILED DESCRIPTION:
This study aims at evaluating the effect from Nephure in reducing dietary oxalate in healthy volunteers on a controlled diet as compared to placebo. Subjects are on a normal diet with controlled oxalate (750mg/day) and calcium (550mg/day) levels for 8 consecutive days. The study is a cross-over design with two four-day treatment periods. The study intends to determine level of reduction in urinary oxalate output as a measure of the effect of Nephure on dietary oxalate when ingested with a meal.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has granted written informed consent.
2. Subject must be a male or non-pregnant female, at least 18 to 55 years of age at the time of Screening, and non-smoker for at least 3 months at the time of screening and throughout study.
3. Subject has a BMI of 18.5 - 29.9 kg/m2 at the time of Screening.
4. Subject has an estimated glomerular filtration rate (eGFR) of >90 mL/min/1.73 m2 at the time of Screening (GFR is calculated using the NIDDK provided equation at the following web address: www.niddk.nih.gov/health-information/communication-programs/nkdep/laboratory-evaluation/glomerular-filtration-rate-calculators/ckd-epi-adults-conventional-units.)
5. Subject has a urinary oxalate <40.5mg/24 hours at the time of Screening .
6. Subject has a urinary uric acid <750mg/24hour at the time of Screening1.
7. Subject is in good health as determined by complete physical examination, medical history, vital signs, and laboratory tests.
8. Subject is able to understand the study and be able to comply to the requirements and restrictions, including agreeing to complete the 24-hour urine collections, and has the ability to report their symptoms.
9. Subject is able to comply with all dietary expectations and fluid intake at the discretion of the Principal Investigator (PI).
10. Female subjects must agree to use an acceptable form of birth control from screening through the duration of the study (unless otherwise stated). See section 5.1.1.

Exclusion Criteria:

1. Subject has a history or presence of clinically significant cardiovascular, pulmonary, respiratory, digestive, hepatic, renal, hematological, gastrointestinal (e.g., active bowel disease, known gallstones, GERD, etc.), endocrine, metabolic, immunological, infectious, dermatologic, neurological, psychological, or psychiatric disease or gastrointestinal surgeries (e.g., bowel resection, gastric bypass, cholecystectomy within the 6 months prior to screening, etc.), in the opinion of the Principal Investigator.
2. Subject has received a positive result for urine drug screen at the screening visit or on Day -3, or has a history of positive test result(s) for human immunodeficiency virus (HIV) antibody, Hepatitis B surface antigen or Hepatitis C antibody.
3. Subject has a history of or a current clinically significant medical condition, allergy, food sensitivity (e.g. maltodextrin) or surgical intervention that might significantly compromise the safety of the subject, interfere with study assessments, or impact the validity of the study results, in the opinion of the Principal Investigator.
4. Subject is taking a medication that would indicate significant anxiety, depression, serious or unstable illness, or lack of good general health, that could interfere with the subject's ability to adhere to study instructions, or complete the study, in the opinion of the Principal Investigator and with approval of the Sponsor.
5. Subject is unable or unwilling to discontinue use of dietary supplements (vitamins, minerals, and/or supplements) throughout the duration of the study or has used these products within 7 days prior to screening.
6. Subject has continuously used (not including intermittent or rare PRN use) prescription or over the counter: proton pump inhibitors within 12 weeks of screening; or H2 blockers within 6 weeks of screening; or antacids within 2 weeks of screening.
7. Subject is currently using medication that could affect oxalate handling such as cholestyramine, any carbonic anhydrase inhibitor, any steroid, any diuretic, any immunosuppressant drug, or has received chemotherapy or systemic immunosuppressive drugs within 6 mos. of their screening visit.
8. Subject has had a clinically significant surgical procedure within 3 mos. prior to the Screening visit or planned surgical procedure during the study conduct.
9. Subject has received an investigational product, device, or therapy within 30 days prior to screening.
10. Subject has been on a self-restricted, controlled, or special therapeutic diet, or has had substantial changes in eating or bowel habits, or have had new GI complaints, within 30 days of their screening visit.
11. Subject has been on systemic antibiotic therapy within 6 weeks prior to the screening visit or plans antibiotic therapy during the study conduct.
12. Subject has a history of allergy or hypersensitivity to the study products, its excipients or any comparable products or excipients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-08-05 (Actual); Study Completion 2018-08-05 (Actual)

PRIMARY OUTCOMES:
Within-Subject Urinary Oxalate Excretion | 8 days
  Milligram of oxalate per 24 hours is determined on dosing days. Within-subject difference in 24 hours urinary oxalate excretion between placebo and Nephure is determined.
Between Groups Urinary Oxalate Excretion | 8 days
  Milligram of oxalate per 24 hours is determined on dosing days. Mean difference in 24 hours urinary oxalate excretion between placebo and Nephure groups is determined.

SECONDARY OUTCOMES:
Urinary Oxalate Excretion Compared to Baseline | 8 days
  Difference in 24 hours urinary oxalate excretion between dosing days and the baseline day immediately preceding is determined.
Adverse Events | 8 days
  Number of participants with adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- QPS Bio-Kinetic Clinical Applications, LLC, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cowley H, Yan Q, Koetzner L, Dolan L, Nordwald E, Cowley AB. In vitro and in vivo safety evaluation of Nephure. Regul Toxicol Pharmacol. 2017 Jun;86:241-252. doi: 10.1016/j.yrtph.2017.03.016. Epub 2017 Mar 18. PMID 28322893
- [Derived] Quintero E, Bird VY, Liu H, Stevens G, Ryan AS, Buzzerd S, Klimberg IW. A Prospective, Double-Blind, Randomized, Placebo-Controlled, Crossover Study Using an Orally Administered Oxalate Decarboxylase (OxDC). Kidney360. 2020 Sep 3;1(11):1284-1290. doi: 10.34067/KID.0001522020. eCollection 2020 Nov 25. PMID 35372879